CLINICAL TRIAL: NCT03317392
Title: A Phase 1/2 Study of Combination Olaparib and Radium-223 in Men With Metastatic Castration-Resistant Prostate Cancer With Bone Metastases (COMRADE)
Brief Title: Testing the Safety of Different Doses of Olaparib Given Radium-223 for Men With Advanced Prostate Cancer With Bone Metastasis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01920; NCI-2017-01920 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10096 (Other: Yale University Cancer Center LAO); 10096 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2017-10-20; First posted 2017-10-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; olaparib; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (radium Ra 223 dichloride, olaparib) (Experimental): Patients receive radium Ra 223 dichloride IV over 1 minute on day 1. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI as well as blood sample collection and a tissue biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Other: Quality-of-Life Assessment; Radiation: Radium Ra 223 Dichloride
- Arm II (radium Ra 223 dichloride) (Experimental): Patients receive radium Ra 223 dichloride as in Arm I. Patients with radiographic progression may crossover to Arm I. If patients have already completed all 6 infusions of radium, they will receive monotherapy with olaparib. If they have not yet completed all 6 radium-223 infusion, they will continue radium-223 infusion until completion and receive concurrent treatment with olaparib. Patients also undergo CT or MRI as well as blood sample collection and a tissue biopsy during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Radiation: Radium Ra 223 Dichloride

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Arm I (radium Ra 223 dichloride, olaparib)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radium Ra 223 Dichloride — Given IV
  Other Names: Alpharadin; BAY 88-8223; BAY88-8223; Radium 223 Dichloride; RADIUM RA-223 DICHLORIDE; Radium-223 Chloride; Radium-223 Dichloride; Xofigo

SUMMARY:
This phase I/II trial studies the best dose and side effects of olaparib and how well it works with radium Ra 223 dichloride in treating patients with castration-resistant prostate cancer that has spread to the bone and other places in the body (metastatic). PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Radioactive drugs, such as radium Ra 223 dichloride, may carry radiation directly to tumor cells and not harm normal cells. Giving olaparib and radium Ra 223 dichloride may help treat patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of olaparib in combination with radium Ra 223 dichloride (radium-223). (Phase 1) II. Evaluate the radiographic progression-free survival (rPFS). (Phase 2)

SECONDARY OBJECTIVES:

I. Evaluate safety and tolerability as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

II. To evaluate rPFS as stratified by disease extent (=< 20 or > 20 bone lesions) and prior docetaxel use (yes or no).

III. Evaluate rPFS in patients harboring or lacking evidence of homologous recombination deficiency (HRD).

IV. Evaluate rPFS in patients based on prior abiraterone and/or next generation androgen receptor (AR) antagonist (enzalutamide, apalutamide, darolutamide or other agent) use (yes versus no) for either hormone sensitive or castration resistant prostate cancer (CRPC).

V. Evaluate prostate specific antigen (PSA) response rate as defined by >= 50% decline in PSA from baseline.

VI. Evaluate total alkaline phosphatase response defined as a reduction of >= 30% from the baseline value, confirmed >= 4 weeks later.

VII. Evaluate time to PSA progression as defined by Prostate Cancer Clinical Trials Working Group (PCTWG) 3 criteria.

VIII. Evaluate radiographic objective response rate as defined by Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1.

IX. Evaluate time to increase in the total alkaline phosphatase (ALP) level defined as an increase of >= 25% from baseline at >= 12 weeks, in patients with no decrease from baseline, or as an increase of >= 25% above the nadir, confirmed >= 3 weeks later, in patients with an initial decrease from baseline.

X. Evaluate time to first subsequent anti-cancer therapy (including AR signaling agents, cytotoxic chemotherapy, immunotherapy, or investigational agents) or death.

XI. Evaluate time to first symptomatic skeletal event (SSE). XII. Evaluate overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Evaluate impact on quality of life (QOL) as determined by Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire and Brief Pain Inventory (BPI).

II. Estimate the frequency of mutations in the deoxyribonucleic acid (DNA) repair pathway in patients with metastatic castration-resistant prostate cancer (CRPC) as determine by Oncopanel testing and by whole exome sequencing (WES).

III. Characterize changes in ribonucleic acid (RNA) expression of DNA repair genes and immune markers by whole transcriptome sequencing (WTS) in each arm.

IV. Characterize changes in immune cell, T-cell receptor (TCR), and B-cell (BCR) receptor repertoire at baseline, during treatment, and at progression in each arm.

V. Evaluate changes in lactate dehydrogenase (LDH) in patients each treatment arm.

VI. Assess the prevalence of germline mutations in homologous recombination genes in all enrolled patients.

VII. Correlate homologous recombination gene germline mutation status with PSA response by treatment arm.

VIII. Evaluate family history of cancers in the study population and correlate family cancer history with germline mutation status.

IX. Correlate presence or absence of RAD51 with somatic and germline homologous recombination gene mutation status, PSA response, and PFS between treatment arms.

X. Evaluate the changes in whole genome sequencing (WGS) of plasma cell-free circulating DNA (cfDNA) based patient-tumor specific signature at baseline, on treatment, and at progression.

XI. Evaluate tumor mutation burden (TMB) and tumor mutational signature in plasma cfDNA at baseline and correlate to tumor tissue TMB and mutational signature.

OUTLINE: This is a phase I, dose-escalation study of olaparib followed by a phase II study.

PHASE I: Patients receive radium Ra 223 dichloride intravenously (IV) over 1 minute on day 1. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive olaparib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) as well as blood sample collection and a tissue biopsy during screening and on study.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive radium Ra 223 dichloride IV over 1 minute on day 1. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI as well as blood sample collection and a tissue biopsy during screening and on study.

ARM II: Patients receive radium Ra 223 dichloride as in Arm I. Patients with radiographic progression may crossover to Arm I. If patients have already completed all 6 infusions of radium, they will receive monotherapy with olaparib. If they have not yet completed all 6 radium-223 infusion, they will continue radium-223 infusion until completion and receive concurrent treatment with olaparib. Patients also undergo CT or MRI as well as blood sample collection and a tissue biopsy during screening and on study.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be male aged >= 18 years of age
* Participants must have histologically or cytologically confirmed adenocarcinoma of the prostate
* Participants must have castrate levels of serum testosterone < 50 ng/dL
* Participants without orchiectomy must be maintained on luteinizing hormone releasing hormone (LHRH) agonist/antagonist; participants receiving prior docetaxel abiraterone, or next generation AR antagonist (enzalutamide, apalutamide, or darolutamide) for hormone sensitive disease are permitted
* Participants must have progressive disease as defined by any of the following:

  * Castrate resistant disease as defined by PCWG-3 criteria; participants must have a rise in PSA on two successive determination at least one week apart and PSA levels >= 2 ng/mL (only the screening PS needs to be >= 2 ng/mL) and serum testosterone < 50 ng/dL
  * Soft tissue progression as defined by RECIST version 1.1
  * Bone disease progression as defined by PCWG-3 criteria including the development of two or more new lesions on bone scan
* Participants must have >= 2 bone metastases by radiographic imaging and at least 1 lesion which has not been treated with prior radiation therapy
* Participants must have tumor accessible for biopsy and be agreeable to baseline tumor biopsy; a metastatic focus is preferred but if not available and prostate is still intact prostate biopsy can be performed
* Availability at the study site of formalin-fixed, paraffin-embedded (FFPE) archival tumor specimens, when available
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* White blood cell count (WBC) >= 3,000/mcL (within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 28 days prior to administration of study treatment)
* Platelets >= 100,000/mcL (within 28 days prior to administration of study treatment)
* Hemoglobin >= 10 g/dL (transfusions permitted) (within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment); for subjects with Gilbert's disease =< 3.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x institutional ULN (within 28 days prior to administration of study treatment)
* Creatinine clearance >= 51 ml/min as defined by Cockcroft-Gault equation (within 28 days prior to administration of study treatment)
* Participants should be receiving an osteoclast targeting agent including either bisphosphonates or denosumab except in patients with contraindications as determined by the treating investigator including:

  * Hypocalcemia
  * Hypophosphatemia
  * Renal impairment including those with a glomerular filtration rate < 35 mL/min using the Cockcroft-Gault equation
  * Hypersensitivity to drug formulation
  * Dental condition or need for dental intervention that per the investigator would increase the risk of osteonecrosis of the jaw
* The effects of olaparib and radium-223 on the developing human fetus are unknown; for this reason, men treated or enrolled on this protocol must agree to use adequate contraception and avoid sperm donation prior to the study, for the duration of study participation, and three months after discontinuation of olaparib and radium-223 administration
* Human immunodeficiency virus (HIV)-positive with negative viral loads on stable antiretroviral regimen and CD4 count > 250 are eligible
* Ability to understand and the willingness to sign a written informed consent document; patients with impaired decision-making who have a legal guardian (e.g., spouse) able to make informed decisions on behalf of the patient are eligible
* Patients must be able to tolerate oral medications by mouth and not have a gastrointestinal illness that would preclude absorption of olaparib

Exclusion Criteria:

* Pathology consistent with small cell carcinoma of the prostate
* Presence of visceral metastases (liver, lung, brain, etc.) or malignant lymphadenopathy exceeding 4 centimeters (cm) in short diameter
* Prior treatment with radium-223
* Prior treatment with olaparib or other PARPi
* Treatment with abiraterone, apalutamide, or darolutamide within 2 weeks of treatment initiation; treatment with cytotoxic chemotherapy within 3 weeks of treatment initiation; treatment with investigational prostate cancer directed therapy within 4 weeks of treatment initiation; treatment with enzalutamide within 4 weeks of treatment initiation
* Prior hemibody external radiotherapy
* Palliative radiation therapy to the bone or other sites within 2 weeks of treatment initiation
* Participants who are receiving any other investigational agents
* Imminent or established spinal cord compression based on clinical and/or imaging findings
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring need for intravenous anti-microbials, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Clinically significant medical condition defined as:

  * Cerebral infarction within 6 months of study treatment
  * Transient ischemic attack within 3 months of study treatment
  * Myocardial infarction within 6 months of study treatment
  * Uncontrolled angina within 3 months of study treatment
  * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or subjects with history of congestive heart failure NYHA class 3 or 4 in the past, or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan performed within 3 months of the screening visit results in a left ventricular ejection fraction that is >= 45%
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes)
  * Prolonged corrected QT interval by the Fridericia correction formula on the screening electrocardiogram (ECG) > 470 msec (as determined on 2 or more time points within a 24 hour period if the first ECG demonstrates a prolonged corrected QT interval) or family history of long QT syndrome
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  * Uncontrolled hypertension as indicated by a resting systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the screening visit
  * History of hypertensive emergency or encephalopathy within 6 months of study treatment
  * Deep venous thrombosis or pulmonary embolism within 3 months of study treatment
* Major surgery within 4 weeks of study treatment; subjects with clinically relevant ongoing complications from prior surgery are not eligible
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Patient unable to swallow orally administered medication
* History of bowel obstruction within 1 month of study treatment
* History of abdominal fistula, intra-abdominal abscess, or gastrointestinal perforation within the 3 months of study treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or radium-223
* Participants receiving strong CYP3A4/5 inducers or inhibitors are ineligible; dihydropyridine calcium-channel blockers are permitted for management of hypertension; the required washout period prior to starting olaparib is 2 weeks for CYP3A inhibitors; the required washout period prior to starting olaparib is 4 weeks for enzalutamide or phenobarbital and 3 weeks for other CYP3A inducers
* Patients with known active hepatitis (i.e. hepatitis B or C) infection
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML
* Patient having received prior allogenic bone marrow transplant or double umbilical cord blood transplantation
* Individuals with a history of a different malignancy are ineligible except for the following circumstances:

  * Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, or
  * Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: superficial bladder cancer, basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of olaparib and radium Ra 223 dichloride | Up to 2 years
Radiographic progression-free survival (rPFS) | Up to 2 years
  Will be estimated using the Kaplan-Meier method by treatment arm. A stratified Cox proportional hazards regression model will estimate the rPFS treatment hazard ratio with 80% 2-sided confidence intervals (CIs).

SECONDARY OUTCOMES:
Radiographic progression free survival (rPFS) | Up to 2 years
  Treatment comparison in rPFS will be conducted in pre-defined subgroups, including homologous recombination deficiency status (yes/no), disease extent (=< 20 or > 20 bone lesions) and prior docetaxel (yes or no). Cox regression hazard ratios (for treatment comparison) along two-sided 80% CI will be provided for each subgroup.
Prostate specific antigen (PSA) response | Up to 2 years
  Will be defined by 50% decline in PSA from baseline. Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Response rate by different criteria will be summarized as number and percentage of participants by treatment arm with two-sided 80% CI and compared between groups using Fisher's exact tests.
Alkaline phosphatase (ALP) response | Up to 2 years
  Will be defined as >= 30% reduction of the blood level, compared to the baseline value. Will be assessed by RECIST 1.1. Response rate by different criteria will be summarized as number and percentage of participants by treatment arm with two-sided 80% CI and compared between groups using Fisher's exact tests.
Tumor response | Up to 2 years
  Will be assessed by RECIST 1.1. Response rate by different criteria will be summarized as number and percentage of participants by treatment arm with two-sided 80% CI and compared between groups using Fisher's exact tests.
Prostate specific antigen (PSA) progression | From randomization to PSA progression by Prostate Cancer Working Group (PCWG) 3 criteria, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms using the stratified log-rank test.
ALP progression | From randomization to the date of first ALP progression, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms using the stratified log-rank test.
Symptomatic skeletal event (SSE) | From randomization to occurrence of the first SSE, such as pathologic bone fracture, spinal cord compression, hypercalcemia of malignancy or radiation therapy or surgery to bone, described by the US Food and Drug Administration, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms using the stratified log-rank test.
Overall survival (OS) | From randomization to the date of death due to any cause, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms using the stratified log-rank test.
Incidence of adverse events | Up to 2 years
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5. Adverse events will be summarized according to grade, overall and by treatment arm, as number and percentage of participants. All adverse events resulting in discontinuation, dose modification, and/or dosing interruption, and/or treatment delay of drug will also be summarized by treatment arm.

OTHER OUTCOMES:
Change in levels of serum lactate dehydrogenase (LDH) | Baseline up to 2 years
  Will be summarized at baseline and each cycle with descriptive statistics. Percent change from baseline or status change (e.g. from normal to abnormal defined by institution upper limit level) will be reported and compared between treatment arms at selected timepoints using Wilcoxon rank sum test or Fisher's exact test as appropriate.
Frequency of mutations in the deoxyribonucleic acid (DNA) repair pathway | Up to 2 years
  Will be determined by Oncopanel testing. Gene mutation frequencies and mean +/- standard deviation of quantitative biomarkers will be summarized by arm and in overall population at baseline and/or at time of progression.
Homologous recombination deficiency | Up to 2 years
  Cox regression or logistic regression will be conducted to explore the association of rPFS or treatment response (PSA or tumor response) with homologous recombination gene mutation status.
Prevalence of germline mutations in homologous recombination genes | Up to 2 years
  Their correlation with family history of cancers as determined by the Family History Questionnaire and PSA response will be evaluated using Fisher's exact test or logistic regression as appropriate in all patients and/or by treatment arm as exploratory analyses.
Quality of life (QOL) | Baseline up to 2 years
  Will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire and Brief Pain Inventory (BPI). For each treatment group, calculated QOL scores will be summarized at baseline and each time point. Changes from baseline will be graphically presented. The effect of treatment will be evaluated using a repeated measures model to incorporate assessments across time into a single analysis, using model contrasts to compare treatment groups at selected time points.

CONTACTS AND LOCATIONS:
Overall Officials: Rana R McKay, Principal Investigator — Yale University Cancer Center LAO
Locations (22):
- United States (22):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm